CLINICAL TRIAL: NCT03530020
Title: Wear Characteristics and Clinical Performance of Lithium Silicate Versus Monolithic Zirconia Crowns. (Randomized Controlled Clinical Trial)
Brief Title: Wear Characteristics and Clinical Performance of Lithium Silicate Versus Monolithic Zirconia Crowns.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rasmia Mamdouh Ali Salem, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: enamel and ceramics wear
Record Dates: First submitted 2018-05-07; First posted 2018-05-21 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2019-01

CONDITIONS: Enamel and Ceramics Wear
Keywords: monolithic zirconia; tooth wear; all ceramic crown
MeSH Terms: conditions — Tooth Wear | interventions — obsidian

STUDY DESIGN:
Intervention Model Description: Patient will receive a restoration with superior function, esthetics, and excellent clinical performance.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- monolithic zirconia crowns (Active Comparator): Monolithic zirconia attracts many dentists worldwide due to its excellent mechanical properties, biocompatibility and appreciate aesthetics
  Interventions: Other: monolithic zirconia crowns
- lithium silicate crowns (Experimental): A lithium silicate glass ceramic is newly introduced to the market. After crystallization, it exhibits an ideal combination of aesthetics and strength with translucency that mirrors the vitality of natural teeth for fabrication of full anatomic anterior and posterior crowns.
  Interventions: Other: lithium silicate crowns

INTERVENTIONS:
Other: monolithic zirconia crowns — full anatomical monolithic crowns
  Other Names: katana zirconia, Kuraray Noritake , Japan
  Arms: monolithic zirconia crowns
Other: lithium silicate crowns — lithium silicate glass ceramics are highly resistance to chipping
  Other Names: obsidian, Glide well Laboratories, USA
  Arms: lithium silicate crowns

SUMMARY:
The aim of the present study is to evaluate the wear characteristics and clinical performance of lithium silicate crowns in comparison to monolithic zirconia crowns.

The quality of the overall restorations as well as gingival tissues will be also evaluated according to modified United States Public Health Service (USPHS) criteria: (Marginal adaptation, color match, anatomic form, integrity of restoration, secondary caries, retention, tooth sensitivity, gingival index and periodontal index) at baseline, 6 months and 1 year

DETAILED DESCRIPTION:
Recently advances in ceramics have greatly improved the mechanical and optical properties of restorative materials to overcome the drawbacks of all ceramic restorations over decades such as fracture, chipping, crack, wear and delamination of veneer ceramics.

Up to date despite the popularity of all ceramic restoration, the clinicians have been worried about the wear of tooth enamel antagonist to ceramic materials.

The wear properties of the ceramic restoration can affect the rate of wear of the antagonist enamel. So the wear resistance of ceramic restoration must be the same as enamel.

Explanation for choice of the comparator:

Monolithic zirconia attracts many dentists worldwide due to its excellent mechanical properties, biocompatibility and appreciate aesthetics. Some in vivo studies demonstrated the clinical success of monolithic zirconia restorations as an antagonist to natural enamel with good marginal adaptation, accepted contour, occlusion and minimum gingival response.

Batson et al. studied the quality of CAD/CAM fabricated single tooth restorations (Ten zirconia restorations were compared to 12 metal ceramic and 10 lithium disilicate counterparts) .They found that were no significant differences between the studied crown systems. No difference of the gingival response among the different crown systems. Eighty percent of zirconia crowns needed no occlusal adjustment; also it showed the least amount of marginal discrepancy.

Lohbauer et al. evaluated the amount of wear on the antagonist occlusal surfaces of clinically placed monolithic zirconia premolar and molar crowns using optical profilometry after 2 years of cementation, they found that the mean volume loss for enamel antagonist contacts (n = 7) was measured to 361 μm and the mean of the maximum vertical loss to 204 μm. The mean volume loss for pure ceramic contacts (n = 10) was measured to 333 μm and the mean of the maximum vertical loss to 145 μm.

Mundhe et al.compared the wear of enamel opposing polished zirconia, glazed metal ceramic crowns and natural enamel as a control, one year after the cementation. They found that the occlusal wear of the antagonistic enamel one year after the cementation of metal ceramic crowns ranged from 69.20 ± 4.10 to 179.70 ± 8.09 μm, whereas, for zirconia crowns, it was from 42.10 ± 4.30 to 127.00 ± 5.03 μm.

Stober et al. reported that after 2 years of cementation of the monolithic zirconia crowns, Mean and maximum vertical loss of enamel in occlusal contact areas caused by monolithic zirconia (46 and 151 μm, respectively) was approximately double that caused by contralateral antagonistic enamel (19-26 and 75-115 μm, respectively).

A lithium silicate glass ceramic (obsidian ceramic) is newly introduced to the market. After crystallization, it exhibits an ideal combination of esthetics and strength with translucency that mirrors the vitality of natural teeth for fabrication of full anatomic anterior and posterior crowns. Obsidian ceramic restorations are highly resistant to chipping unlike other ceramics, due to their monolithic composition and average flexural strength of 385 MPa. Also Obsidian Milling Block owes its good wear resistance due to a very high content of ultrafine nanometer-size crystalline structure.

ELIGIBILITY:
Inclusion Criteria:

* All subjects are required to be:

  1. Age range of the patients from 21-50 years old; able to read and sign the informed consent document, illiterate patient will be avoided.
  2. Patients able physically and psychologically to tolerate conventional restorative procedures.
  3. Patients with no active periodontal or pulpal diseases, having teeth with good restorations.
  4. Patients with teeth problems indicated for full coverage restoration (e.g. moderate to severe discoloration, coronal fracture where partial coverage would lack retention, malposed or malformed teeth).
  5. Patients with root canal treated teeth requiring full coverage restorations.
  6. Presence of an opposing natural tooth which is non-restored or minimally restored. (Minimally restored is defined as teeth which have no restoration greater than a Class II a restoration)
  7. The opposing arch doesn't have a full coverage restoration or a partial denture.
  8. Patients willing to return for follow-up examinations and evaluation.

     Exclusion Criteria:

  <!-- -->

  1. Patients with poor oral hygiene.
  2. Patients with psychiatric problems or unrealistic expectation (patient that has phobia from dental treatments or needle bunch).
  3. Patients have no opposite occluding dentition in the area intended for restoration
  4. Patients suffer from Para functional habits or temporomandibular disorders. (as those patient may have wear which will affect the results)

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
Wear of all ceramic crowns and color matching | 12 month
  (Wear of ceramic crowns) of the two groups will be assessed using the 3D optical profilometer.
color matching | 12 month
  Color match of the two groups will assessed using the modified United States public health service (USPHS) criteria as follows:
  * Alpha (Excellent) ideal.
  * Bravo (Acceptable) less than ideal but no modifications required
  * Charlie (Acceptable but modifications needed) staining or other shade modifications required.
  * Delta (Unacceptable) remake.

SECONDARY OUTCOMES:
Wear of enamel antagonist to all ceramic crowns | 12 month
  wear of antagonist enamel of the two groups will be assessed using the 3D optical profilometer.
Marginal adaptation | 12 month
  of the two groups will assessed using the modified United States public health service (USPHS) criteria as follows:
  * Alpha (Excellent) ideal.
  * Bravo (Acceptable) less than ideal but no modifications required
  * Charlie (Acceptable but modifications needed) modifications required.
  * Delta (Unacceptable) remake.
anatomic form | 12 month
  of the two groups will assessed using the modified United States public health service (USPHS) criteria as follows:
  * Alpha (Excellent) ideal.
  * Bravo (Acceptable) less than ideal but no modifications required
  * Charlie (Acceptable but modifications needed) modifications required.
  * Delta (Unacceptable) remake.
integrity of restoration | 12 month
  of the two groups will assessed using the modified United States public health service (USPHS) criteria as follows:
  * Alpha (Excellent) ideal.
  * Bravo (Acceptable) less than ideal but no modifications required
  * Charlie (Acceptable but modifications needed) modifications required.
  * Delta (Unacceptable) remake.
secondary caries | 12 month
  of the two groups will assessed using the modified United States public health service (USPHS) criteria as follows:
  * Alpha (Excellent) ideal.
  * Bravo (Acceptable) less than ideal but no modifications required
  * Charlie (Acceptable but modifications needed) modifications required.
  * Delta (Unacceptable) remake.
retention | 12 month
  of the two groups will assessed using the modified United States public health service (USPHS) criteria as follows:
  * Alpha (Excellent) ideal.
  * Bravo (Acceptable) less than ideal but no modifications required
  * Charlie (Acceptable but modifications needed) modifications required.
  * Delta (Unacceptable) remake.
opposing tooth sensitivity | 12 month
  of the two groups will assessed using the modified United States public health service (USPHS) criteria as follows:
  * Alpha (Excellent) ideal.
  * Bravo (Acceptable) less than ideal but no modifications required
  * Charlie (Acceptable but modifications needed) modifications required.
  * Delta (Unacceptable) remake.
gingival condition | 12 month
  Gingival index by Visual inspection using Score from 0-3
periodontal condition | 12 month
  Periodontal index by Periodontal probe using Score from 0-4

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Giza, Egypt

REFERENCES:
- [Background] Larsson C, Wennerberg A. The clinical success of zirconia-based crowns: a systematic review. Int J Prosthodont. 2014 Jan-Feb;27(1):33-43. doi: 10.11607/ijp.3647. PMID 24392475
- [Background] Daou EE. Esthetic Prosthetic Restorations: Reliability and Effects on Antagonist Dentition. Open Dent J. 2015 Dec 31;9:473-81. doi: 10.2174/1874210601509010473. eCollection 2015. PMID 26962376
- [Background] Mehta SB, Banerji S, Millar BJ, Suarez-Feito JM. Current concepts on the management of tooth wear: part 1. Assessment, treatment planning and strategies for the prevention and the passive management of tooth wear. Br Dent J. 2012 Jan 13;212(1):17-27. doi: 10.1038/sj.bdj.2011.1099. PMID 22240686
- [Background] Mundhe K, Jain V, Pruthi G, Shah N. Clinical study to evaluate the wear of natural enamel antagonist to zirconia and metal ceramic crowns. J Prosthet Dent. 2015 Sep;114(3):358-63. doi: 10.1016/j.prosdent.2015.03.001. Epub 2015 May 16. PMID 25985742
- [Background] Olivera AB, Marques MM. Esthetic restorative materials and opposing enamel wear. Oper Dent. 2008 May-Jun;33(3):332-7. doi: 10.2341/07-95. PMID 18505225
- [Background] Magne P, Oh WS, Pintado MR, DeLong R. Wear of enamel and veneering ceramics after laboratory and chairside finishing procedures. J Prosthet Dent. 1999 Dec;82(6):669-79. doi: 10.1016/s0022-3913(99)70008-9. PMID 10588803
- [Background] Burgess JO, Janyavula S, Lawson NC, Lucas TJ, Cakir D. Enamel wear opposing polished and aged zirconia. Oper Dent. 2014 Mar-Apr;39(2):189-94. doi: 10.2341/12-345-L. Epub 2013 Jul 12. PMID 23848069
- [Background] Preis V, Weiser F, Handel G, Rosentritt M. Wear performance of monolithic dental ceramics with different surface treatments. Quintessence Int. 2013 May;44(5):393-405. doi: 10.3290/j.qi.a29151. PMID 23479579
- [Background] Park JH, Park S, Lee K, Yun KD, Lim HP. Antagonist wear of three CAD/CAM anatomic contour zirconia ceramics. J Prosthet Dent. 2014 Jan;111(1):20-9. doi: 10.1016/j.prosdent.2013.06.002. Epub 2013 Nov 5. PMID 24199603
- [Background] Janyavula S, Lawson N, Cakir D, Beck P, Ramp LC, Burgess JO. The wear of polished and glazed zirconia against enamel. J Prosthet Dent. 2013 Jan;109(1):22-9. doi: 10.1016/S0022-3913(13)60005-0. PMID 23328193
- [Background] Stober T, Bermejo JL, Rammelsberg P, Schmitter M. Enamel wear caused by monolithic zirconia crowns after 6 months of clinical use. J Oral Rehabil. 2014 Apr;41(4):314-22. doi: 10.1111/joor.12139. Epub 2014 Jan 22. PMID 24447258
- [Background] Lawson NC, Janyavula S, Syklawer S, McLaren EA, Burgess JO. Wear of enamel opposing zirconia and lithium disilicate after adjustment, polishing and glazing. J Dent. 2014 Dec;42(12):1586-91. doi: 10.1016/j.jdent.2014.09.008. Epub 2014 Sep 23. PMID 25257823
- [Background] Samer MS, Faraz Q, Al-Dubai SAR, Vohra F, Abdullah H, Taiyeb-Ali TB, Saub R. Clinical Outcomes and Predictors of Satisfaction in Patients with Improved Lithium Disilicate All-Ceramic Crowns. Med Princ Pract. 2017;26(5):470-479. doi: 10.1159/000481864. Epub 2017 Oct 1. PMID 28965115
- [Background] Cvar JF, Ryge G. Reprint of criteria for the clinical evaluation of dental restorative materials. 1971. Clin Oral Investig. 2005 Dec;9(4):215-32. doi: 10.1007/s00784-005-0018-z. No abstract available. PMID 16315023
- [Background] Lohbauer U, Reich S. Antagonist wear of monolithic zirconia crowns after 2 years. Clin Oral Investig. 2017 May;21(4):1165-1172. doi: 10.1007/s00784-016-1872-6. Epub 2016 Jun 9. PMID 27277661
- [Background] Suputtamongkol K, Anusavice KJ, Suchatlampong C, Sithiamnuai P, Tulapornchai C. Clinical performance and wear characteristics of veneered lithia-disilicate-based ceramic crowns. Dent Mater. 2008 May;24(5):667-73. doi: 10.1016/j.dental.2007.06.033. Epub 2007 Aug 28. PMID 17727943
- [Background] Batson ER, Cooper LF, Duqum I, Mendonca G. Clinical outcomes of three different crown systems with CAD/CAM technology. J Prosthet Dent. 2014 Oct;112(4):770-7. doi: 10.1016/j.prosdent.2014.05.002. Epub 2014 Jun 28. PMID 24980739
- [Background] Stober T, Bermejo JL, Schwindling FS, Schmitter M. Clinical assessment of enamel wear caused by monolithic zirconia crowns. J Oral Rehabil. 2016 Aug;43(8):621-9. doi: 10.1111/joor.12409. Epub 2016 May 20. PMID 27198539
- [Background] Landry RG, Jean M. Periodontal Screening and Recording (PSR) Index: precursors, utility and limitations in a clinical setting. Int Dent J. 2002 Feb;52(1):35-40. doi: 10.1111/j.1875-595x.2002.tb00595.x. PMID 11931220